CLINICAL TRIAL: NCT04919486
Title: Investigating the Impacts of Visual Feedback Non-weight Bearing Exercise on Muscle Strength and Physical Fitness of Lower Limbs in Elderly People With Knee Osteoarthritis in the Community.
Brief Title: Visual Feedback Non-weight Bearing Exercise on the Elderly With Knee Osteoarthritis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: N201908020
Record Dates: First submitted 2020-07-29; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2020-07

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Feedback, Sensory

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment group (Experimental): non-weight bearing visual feedback intervention under the of Labview software, and used rowing machine equipment for exercise training for 30 minutes,then eselastic band exercise training for 30 minutes.
  Interventions: Behavioral: visual feedback with non-weight bearing exercise
- elastic band exercise (Active Comparator): elastic band exercise under the Physiotherapist, and used elastic band for exercise training for 60 minutes,include muscles flexion the hip joint, muscles extention the hip joint,etc.
  Interventions: Behavioral: elastic band exercise

INTERVENTIONS:
Behavioral: visual feedback with non-weight bearing exercise — the training time is 12 weeks, twice a week, 60 minutes each time, a total of 24 times.
  Arms: Experiment group
Behavioral: elastic band exercise — the training time is 12 weeks, twice a week, 60 minutes each time, a total of 24 times.
  Arms: elastic band exercise

SUMMARY:
Degenerative knee arthritis is the most common chronic arthritis disease. Once the elderly suffer from this disease, it will accelerate the loss of body function and autonomy. strength performances and maintain are the most important functional performances of lower extremities, especially in walking and balance in daily activities for elderly people with osteoarthritis(OA) of the knee. However, combining the exercise and visual feedback may promote the muscle strength and functional performances of lower limbs, facilitating the muscle strength, motor and boady functional performances for elderly adults after OA knee. Therefore, the purpose of this proposal is to investigate the changes in muscle strength and physical fitness of lower limbs in older adults following OA knee after visual feedback non-weight bearing exercise intervention.

DETAILED DESCRIPTION:
Backgroud:In clinical observation, aging leads to a gradual degeneration of the neuromuscular system, decreasing the muscle strength and functional performances of lower extremities. Muscle strength performances and maintain are the most important functional performances of lower extremities, especially in walking and balance in daily activities for elderly people with osteoarthritis(OA) of the knee. However, non-weight bearing exercise combing visual feedback may promote functional performances of lower limbs, facilitating the muscle strength for elderly people with OA knee.

Purpose: Therefore, the purpose of this proposal is to promote muscle strength and physical fitness after visual feedback non-weight bearing exercise intervention.

Method:After recruiting 40 elderly people with degenerative knee arthritis, they were randomly assigned to the experimental group and the control group .The experimental group conducted visual feedback under the guidance of Labview software, and used rowing machine equipment for resistance exercise training.The training time of the two groups is 12 weeks, twice a week, 30 minutes each time, a total of 24 times.Before and after exercise training , both groups used the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) to understand their self-response of knee(pain、stiffness functional)；used MicroFets3 to measure hip and knee muscle strength；Elder Functional Fitness chose Chair stand test、Functional reach test、10m-Walking time are used to understand the body function.

Stastistical analysis:Data were analyzed with SPSS18.0. Paired Sample t-test and Independent-Sample T Test were used to determine the between-groupand within-group differences on all outcome measures. The statistical significance level was set at a (p<0.05).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of degenerative knee arthritis.
* Must be able to stand up and sit down.

Exclusion Criteria:

* surgery on the knee or hip joint.
* rheumatoid arthritis and uarthritis in past six years.
* lower limb fractures
* neurological diseases,e.g.,stroke、parkinson's disease
* injected hyaluronic acid into the knee joint in the past two months
* severe cardiovascular and heart failure.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-07-25 (Actual); Primary Completion 2021-07-25 (Estimated); Study Completion 2021-07-25 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 5 minutes
  The scale is mainly to trace the patient's subjective perception of the knee joint within 48 hours. There are 24 questions, divided into three aspects: pain (5 questions, 0-20 points), stiffness (2 questions, 0-8 points) , Functional activities (17 questions, 0-68 points), each item is divided into five levels: none, minor, moderate, severe, and very severe. The total of the three parts is 0-96 points.

SECONDARY OUTCOMES:
MicroFets3 to measure hip and knee muscle strength | 20 minutes
  we Include Hip Abductor 、Hip adductors、Hip extensors、Hip flexors、knee extensors、knee flexors etc.Before the test, the subject practiced once and then performed a formal test. The strength of each muscle contraction was recorded in kilograms. During the formal test, the subject was required to resist MicroFET3 with maximum strength, and the tester gave the order (Strong! Push hard! Push hard!), the data uses the average of three times, and each muscle rests for one minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei, Taipei, Taiwan

REFERENCES:
- [Derived] Lin PL, Yu LF, Kuo SF, Wang XM, Lu LH, Lin CH. Effects of computer-aided rowing exercise systems on improving muscle strength and function in older adults with mild knee osteoarthritis: a randomized controlled clinical trial. BMC Geriatr. 2022 Oct 21;22(1):809. doi: 10.1186/s12877-022-03498-2. PMID 36266615